CLINICAL TRIAL: NCT01395966
Title: Clinical Study to Assess the Efficacy and Safety of DF289 Plus DF277 Otic Solution in the Treatment of Middle Ear Infections in Pediatric Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Salvat (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DF289III/10IA02
Record Dates: First submitted 2011-07-08; First posted 2011-07-18 (Estimated); Results first posted 2015-10-22 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-09

CONDITIONS: Acute Otitis Media
Keywords: with tubes
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- DF289 (Active Comparator): Ear drops
  Interventions: Drug: DF289
- DF277 (Active Comparator): Ear drops
  Interventions: Drug: DF277
- DF289 plus DF277 (Experimental): Ear drops
  Interventions: Drug: DF289 plus DF277

INTERVENTIONS:
Drug: DF289 — Ear drops
  Arms: DF289
Drug: DF277 — Ear drops
  Arms: DF277
Drug: DF289 plus DF277 — Ear drops
  Arms: DF289 plus DF277

SUMMARY:
The purpose of this study is to determine if the combination of DF289 plus DF277 is safe and effective in treating middle ear infections in children with ear tubes.

ELIGIBILITY:
Inclusion Criteria:

* 6 months to 12 years
* ear tube in the ear which will be treated
* otorrhea for 3 weeks or less
* moderate or severe otorrhea

Exclusion Criteria:

* other ear diseases

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 331 (Actual)
Dates: Start 2011-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratorios Salvat, S.A., Esplugues de Llobregat, Barcelona, Spain

REFERENCES:
- [Derived] Spektor Z, Pumarola F, Ismail K, Lanier B, Hussain I, Ansley J, Butehorn HF 3rd, Esterhuizen K, Byers J, Douglis F, Lansford B, Hernandez FJ. Efficacy and Safety of Ciprofloxacin Plus Fluocinolone in Otitis Media With Tympanostomy Tubes in Pediatric Patients: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2017 Apr 1;143(4):341-349. doi: 10.1001/jamaoto.2016.3537. PMID 28006041

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DF289 | DF277 | DF289 Plus DF277
Started | 109 | 110 | 112
Completed | 99 | 91 | 104
Not Completed | 10 | 19 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DF289 | DF277 | DF289 Plus DF277 | Total
Number analyzed (Participants) | 109 | 110 | 112 | 331
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 109 | 110 | 112 | 331
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.5 (2.7) | 3.5 (2.6) | 3.2 (2.5) | 3.4 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 68 | 64 | 198
  Male | 43 | 42 | 48 | 133

OUTCOME MEASURES:

1. Primary Outcome: Time to Cessation of Otorrhea
Time Frame: From baseline until the end of the study ( up to 22 days)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | DF289 | DF277 | DF289 Plus DF277
Number analyzed (Participants) | 109 | 110 | 112
days | 7.69 [4.78 to 11.44] | 22 [7.43 to 22] | 3.75 [3.04 to 4.39]

ADVERSE EVENTS:
Time Frame: During all the study (22 days)
Description: Only related TEAE are reported. There were 331 patients randomized, but only 327 were dosed. Only dosed patients are considered for the AE Reporting.
  One patient was randomized to receive DF277 but began taking DF289 Plus DF277. This patient is included in the safety population under DF289 Plus DF277 treatment.
Arm/Group | DF289 | DF277 | DF289 Plus DF277
Serious Adverse Events (participants affected / at risk) | 0/108 | 0/106 | 0/113
Other Adverse Events (participants affected / at risk) | 4/108 | 9/106 | 7/113
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DF289 (N=108) | DF277 (N=106) | DF289 Plus DF277 (N=113)
auricular swelling (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
ear pain (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 1 (1)
otorrhoea (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
ear canal erythema (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
ear haemorrahage (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
otitis media (Infections and infestations) | 1 (1) | 3 (3) | 2 (2)
otitis media acute (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
ear infection fungal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
excessive granulation tissue (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
rash (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor does not object to publication by Institution of the results of the Trial based on information collected or generated by Institution, whether or not the results are favorable to the Sponsor Drug. However, to ensure against inadvertent disclosure of Confidential Information or unprotected Inventions, Institution will provide Sponsor an opportunity to review any proposed publication or other type of disclosure before it is submitted or otherwise disclosed.